CLINICAL TRIAL: NCT02488759
Title: Non-Comparative, Open-Label, Multiple Cohort, Phase 1/2 Study of Nivolumab Monotherapy and Nivolumab Combination Therapy in Subjects With Virus-Positive and Virus-Negative Solid Tumors
Brief Title: An Investigational Immuno-therapy Study to Investigate the Safety and Effectiveness of Nivolumab, and Nivolumab Combination Therapy in Virus-associated Tumors
Acronym: CheckMate358
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-358; 2015-000230-29 (EudraCT Number)
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Results first posted 2022-04-12 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Various Advanced Cancer
MeSH Terms: interventions — Nivolumab; Ipilimumab; relatlimab; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Neoadjuvant Cohort (Experimental): Nivolumab intravenous infusion as specified
  **Not participating: Japan, Korea, and Taiwan
  Interventions: Drug: Nivolumab
- Metastatic Monotherapy Cohort (Experimental): Nivolumab intravenous infusion as specified
  Interventions: Drug: Nivolumab
- Nivolumab plus Ipilimumab Cohort (Experimental): Nivolumab intravenous infusion as specified with Ipilimumab intravenous infusion as specified
  **Not participating: Belgium, France and Germany
  Cohort expansion participating countries: Spain, US, UK, Netherlands, Japan and Mexico
  **Not participating in cohort expansion: France, Germany, Korea and Taiwan
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Nivolumab plus Relatlimab Cohort (Experimental): Nivolumab intravenous infusion as specified with Relatlimab intravenous infusion as specified
  ** Not Participating: Belgium, Germany, France, Japan, Korea, Taiwan, UK, and Netherlands
  Enrollment is closed for this cohort
  Interventions: Drug: Nivolumab; Drug: Relatlimab
- Nivolumab plus Daratumumab Cohort (Experimental): Nivolumab intravenous infusion as specified with Daratumumab intravenous infusion as specified
  **Not Participating: Belgium, Germany, France, Japan, Korea, Taiwan, UK, and Netherlands
  Enrollment is closed for this cohort
  Interventions: Drug: Nivolumab; Drug: Daratumumab

INTERVENTIONS:
Drug: Nivolumab
Drug: Ipilimumab
  Arms: Nivolumab plus Ipilimumab Cohort
Drug: Relatlimab
  Other Names: BMS-986016; Anti-LAG 3
  Arms: Nivolumab plus Relatlimab Cohort
Drug: Daratumumab
  Other Names: Darzalex
  Arms: Nivolumab plus Daratumumab Cohort

SUMMARY:
The purpose of this study to investigate the safety and effectiveness of nivolumab, and nivolumab combination therapy, to treat patients who have virus-associated tumors. Certain viruses have been known to play a role in tumor formation and growth. This study will investigate the effects of the study drugs, in patients who have the following types of tumors:

* Anal canal cancer-No longer enrolling this tumor type
* Cervical cancer
* Epstein Barr Virus (EBV) positive gastric cancer-No longer enrolling this tumor type
* Merkel Cell Cancer
* Penile cancer-No longer enrolling this tumor type
* Vaginal and vulvar cancer-No longer enrolling this tumor type
* Nasopharyngeal Cancer - No longer enrolling this tumor type
* Head and Neck Cancer - No longer enrolling this tumor type

ELIGIBILITY:
Inclusion Criteria:

* Histopathologic confirmation of the following tumor types (please refer to protocol for full details pertaining to eligible tumor types):

  1. Merkel Cell Carcinoma
  2. Gastric or Gastro-Esophageal junction carcinoma (No longer enrolling this tumor type)
  3. Nasopharyngeal Carcinoma
  4. Squamous cell carcinoma (SCC) of the cervix, vagina, or vulva
  5. Squamous cell carcinoma of the Head and Neck
  6. Squamous cell carcinoma of the anal canal and penis
  7. Recurrent/metastatic SCC of the cervix not amenable to curative treatment with surgery and/or radiation therapy who are unsuitable for platinum-based therapy may enroll in the cervical cancer Combination B expansion cohort
* Measurable disease by CT or MRI
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patient willing to comply to provide tumor tissue (archival or fresh biopsy specimen)
* Men and women of age 18 or older

Exclusion Criteria:

* Active brain metastases or leptomeningeal metastases
* Patients with active, known or suspected autoimmune disease
* Patients with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications
* Patients with hepatitis
* Patients with HIV
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2022-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (40):
- United States (14):
  - Local Institution - 0033, Tampa, Florida
  - Local Institution - 0003, Atlanta, Georgia
  - Local Institution - 0023, Lutherville, Maryland
  - Local Institution - 0002, Boston, Massachusetts
  - Local Institution - 0019, Boston, Massachusetts
  - Local Institution - 0020, Boston, Massachusetts
  - Local Institution - 0035, Ann Arbor, Michigan
  - Local Institution - 0036, New York, New York
  - Local Institution - 0022, Charlotte, North Carolina
  - Local Institution - 0005, Oklahoma City, Oklahoma
  - Local Institution - 0004, Portland, Oregon
  - Local Institution - 0029, Pittsburgh, Pennsylvania
  - Local Institution - 0001, Sioux Falls, South Dakota
  - Local Institution - 0021, Seattle, Washington
- Belgium (3):
  - Local Institution - 0012, Brussels
  - Local Institution - 0014, Brussels
  - Local Institution - 0013, Brussels
- France (4):
  - Local Institution - 0031, Marseille
  - Local Institution - 0038, Paris
  - Local Institution - 0032, Toulouse
  - Local Institution - 0030, Vlllejuif
- Germany (2):
  - Local Institution - 0027, Essen
  - Local Institution - 0028, Heilbronn
- Japan (3):
  - Local Institution - 0039, Kashiwa-shi, Chiba
  - Local Institution - 0040, Chuo-ku, Tokyo
  - Local Institution - 0041, Koto-ku, Tokyo
- Mexico (3):
  - Local Institution - 0056, Mexico City, Mexico City
  - Local Institution, Oaxaca City, Oaxaca
  - Local Institution - 0046, Mérida, Yucatán
- Netherlands (2):
  - Local Institution - 0011, Amsterdam
  - Local Institution - 0034, Utrecht
- Local Institution - 0024, Seoul, South Korea
- Spain (3):
  - Local Institution - 0018, Barcelona
  - Local Institution - 0017, Madrid
  - Local Institution - 0016, Navarra
- Taiwan (2):
  - Local Institution - 0037, Tainan
  - Local Institution - 0026, Taipei
- United Kingdom (3):
  - Local Institution - 0006, Glasgow, Lanarkshire
  - Local Institution - 0010, Birmingham, West Midlands
  - Local Institution - 0008, London

REFERENCES:
- [Derived] Bhatia S, Topalian SL, Sharfman W, Meyer T, Steven N, Lao CD, Farinas-Madrid L, Devriese LA, Moore K, Ferris RL, Honma Y, Elias I, Srirangam A, Garnett-Benson C, Lee M, Nghiem P. Nivolumab With or Without Ipilimumab in Patients With Recurrent or Metastatic Merkel Cell Carcinoma: A Nonrandomized, Open-Label, International, Multicenter Phase I/II Study. J Clin Oncol. 2025 Mar 20;43(9):1137-1147. doi: 10.1200/JCO-24-02138. Epub 2025 Jan 31. PMID 39889250
- [Derived] Oaknin A, Moore K, Meyer T, Lopez-Picazo Gonzalez J, Devriese LA, Amin A, Lao CD, Boni V, Sharfman WH, Park JC, Tahara M, Topalian SL, Magallanes M, Molina Alavez A, Khan TA, Copigneaux C, Lee M, Garnett-Benson C, Wang X, Naumann RW. Nivolumab with or without ipilimumab in patients with recurrent or metastatic cervical cancer (CheckMate 358): a phase 1-2, open-label, multicohort trial. Lancet Oncol. 2024 May;25(5):588-602. doi: 10.1016/S1470-2045(24)00088-3. Epub 2024 Apr 9. PMID 38608691
- [Derived] Pulliam T, Jani S, Jing L, Ryu H, Jojic A, Shasha C, Zhang J, Kulikauskas R, Church C, Garnett-Benson C, Gooley T, Chapuis A, Paulson K, Smith KN, Pardoll DM, Newell EW, Koelle DM, Topalian SL, Nghiem P. Circulating cancer-specific CD8 T cell frequency is associated with response to PD-1 blockade in Merkel cell carcinoma. Cell Rep Med. 2024 Feb 20;5(2):101412. doi: 10.1016/j.xcrm.2024.101412. Epub 2024 Feb 10. PMID 38340723
- [Derived] Ferris RL, Spanos WC, Leidner R, Goncalves A, Martens UM, Kyi C, Sharfman W, Chung CH, Devriese LA, Gauthier H, Chiosea SI, Vujanovic L, Taube JM, Stein JE, Li J, Li B, Chen T, Barrows A, Topalian SL. Neoadjuvant nivolumab for patients with resectable HPV-positive and HPV-negative squamous cell carcinomas of the head and neck in the CheckMate 358 trial. J Immunother Cancer. 2021 Jun;9(6):e002568. doi: 10.1136/jitc-2021-002568. PMID 34083421
- [Derived] Topalian SL, Bhatia S, Amin A, Kudchadkar RR, Sharfman WH, Lebbe C, Delord JP, Dunn LA, Shinohara MM, Kulikauskas R, Chung CH, Martens UM, Ferris RL, Stein JE, Engle EL, Devriese LA, Lao CD, Gu J, Li B, Chen T, Barrows A, Horvath A, Taube JM, Nghiem P. Neoadjuvant Nivolumab for Patients With Resectable Merkel Cell Carcinoma in the CheckMate 358 Trial. J Clin Oncol. 2020 Aug 1;38(22):2476-2487. doi: 10.1200/JCO.20.00201. Epub 2020 Apr 23. PMID 32324435
- [Derived] Naumann RW, Hollebecque A, Meyer T, Devlin MJ, Oaknin A, Kerger J, Lopez-Picazo JM, Machiels JP, Delord JP, Evans TRJ, Boni V, Calvo E, Topalian SL, Chen T, Soumaoro I, Li B, Gu J, Zwirtes R, Moore KN. Safety and Efficacy of Nivolumab Monotherapy in Recurrent or Metastatic Cervical, Vaginal, or Vulvar Carcinoma: Results From the Phase I/II CheckMate 358 Trial. J Clin Oncol. 2019 Nov 1;37(31):2825-2834. doi: 10.1200/JCO.19.00739. Epub 2019 Sep 5. PMID 31487218
- [Derived] Appelbaum J, Wells D, Hiatt JB, Steinbach G, Stewart FM, Thomas H, Nghiem P, Kapur RP, Thompson JA, Bhatia S. Fatal enteric plexus neuropathy after one dose of ipilimumab plus nivolumab: a case report. J Immunother Cancer. 2018 Aug 31;6(1):82. doi: 10.1186/s40425-018-0396-9. PMID 30170630
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 578 participants treated
Groups:
- Metastatic Monotherapy: Nivolumab IV over 30 minutes at 240 mg every 2 weeks for a maximum of 24 months or until disease progression, unacceptable toxicity, or withdrawal of consent, whichever comes first
- Metastatic Combo A: Nivolumab 3 mg/kg IV over 30 minutes every 2 weeks + Ipilimumab 1 mg/kg IV over 30 minutes every 6 weeks for a maximum of 24 months or until disease progression, unacceptable toxicity, or withdrawal of consent, whichever comes first
- Metastatic Combo B: Nivolumab 1 mg/kg IV over 30 minutes + Ipilimumab 3 mg/kg IV over 30 minutes every 3 weeks for 4 doses followed by Nivolumab 240 mg IV over 30 minutes every 2 weeks for a maximum of 24 months or until disease progression, unacceptable toxicity, or withdrawal of consent, whichever comes first
- Metastatic Combo C: Nivolumab 240 mg IV over 30 minutes + BMS-986016 (Relatlimab) 80 mg IV over 60 minutes administered every 2 weeks for a maximum of 24 months, or until disease progression, unacceptable toxicity, or withdrawal of consent, whichever comes first
- Metastatic Combo D: Daratumumab 16 mg/kg IV weekly for the first 8 weeks. Starting at Week 3, Nivolumab 240 mg IV over 30 minutes every 2 weeks. Daratumumab 16 mg/kg every 2 weeks from Weeks 9-24. Starting at Week 25, Nivolumab 480 mg IV flat dose over 30 minutes every 4 weeks; daratumumab 16 mg/kg every 4 weeks for a maximum of 24 months or until progression, unacceptable toxicity, or withdrawal of consent, whichever comes first
- Neoadjuvant: Nivolumab administered intravenously (IV) over 30 minutes at 240 mg for 2 doses, on Day 1 and Day 15
Period: Overall Study
Arm/Group | Metastatic Monotherapy | Metastatic Combo A | Metastatic Combo B | Metastatic Combo C | Metastatic Combo D | Neoadjuvant
Started (Started = treated) | 113 | 195 | 133 | 8 | 6 | 123
Completed (Completed = completed the treatment period) | 0 | 0 | 0 | 0 | 0 | 116
Not Completed | 113 | 195 | 133 | 8 | 6 | 7
Not completed — Disease progression | 73 | 111 | 62 | 7 | 4 | 2
Not completed — Study drug toxicity | 11 | 33 | 31 | 0 | 0 | 2
Not completed — Adverse event unrelated to study drug | 9 | 11 | 7 | 0 | 1 | 0
Not completed — Participant request to discontinue study treatment | 6 | 8 | 4 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 3 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Maximum clinical benefit | 3 | 0 | 1 | 0 | 0 | 0
Not completed — Other reasons | 7 | 32 | 23 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metastatic Monotherapy | Metastatic Combo A | Metastatic Combo B | Metastatic Combo C | Metastatic Combo D | Neoadjuvant | Total
Number analyzed (Participants) | 113 | 195 | 133 | 8 | 6 | 123 | 578
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.4 (13.5) | 57.5 (13.2) | 48.2 (12.3) | 59.0 (7.6) | 66.5 (15.3) | 62.0 (12.7) | 56.4 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 85 | 129 | 1 | 3 | 59 | 316
  Male | 74 | 110 | 4 | 7 | 3 | 64 | 262
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2 | 0 | 0 | 2 | 6
  Asian | 14 | 31 | 10 | 0 | 0 | 1 | 56
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 6 | 5 | 0 | 0 | 3 | 17
  White | 86 | 147 | 115 | 8 | 6 | 113 | 475
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 11 | 1 | 0 | 0 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Neoadjuvant: Number of Participants With Drug-Related Select Adverse Events (AEs)
Description: Number of participants with any grade of drug-related select adverse events (AEs) including endocrine, gastrointestinal, hepatic, pulmonary, renal, skin, and hypersensitivity AEs in Neoadjuvant cohort
Time Frame: From first dose to 30 days post last dose (Up to 2 months)
Population: All treated participants in the neoadjuvant cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant
Number analyzed (Participants) | 123
Participants
  Endocrine AEs | 3
  Gastrointestinal AEs | 4
  Hepatic AEs | 3
  Pulmonary AEs | 0
  Renal AEs | 0
  Skin AEs | 9
  Hypersensitivity/Infusion Reaction AEs | 5

2. Primary Outcome: Neoadjuvant: Number of Participants With Drug-Related Serious Adverse Events (SAEs)
Description: Number of participants with any grade of drug-related serious adverse events (SAEs) in Neoadjuvant cohort
Time Frame: From first dose to 30 days post last dose (Up to 2 months)
Population: All treated participants in the neoadjuvant cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant
Number analyzed (Participants) | 123
Participants | 6

3. Primary Outcome: Neoadjuvant: Rate of Surgery Delay
Description: Rate of surgery delay is defined as the percentage of participants in the neoadjuvant cohort with surgery delayed > 4 weeks from the planned surgery date or planned start date for chemoradiation due to a drug-related adverse event.
  Participants with the following diseases will be assessed:
  1. HPV positive squamous cell carcinoma of the Head and Neck (SCCHN);
  2. HPV negative SCCHN;
  3. Cervical Carcinoma;
  4. Vaginal/Vulvar Carcinoma;
  5. Merkel Cell Carcinoma
Time Frame: Day 29
Population: All tumor reduction evaluable participants in the neoadjuvant cohort
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Neoadjuvant
Number analyzed (Participants) | 112
Percentage of participants
  HPV positive SCCHN: number analyzed (Participants) | 25
  HPV positive SCCHN | 0 [0 to 13.7]
  HPV negative SCCHN: number analyzed (Participants) | 25
  HPV negative SCCHN | 0 [0 to 13.7]
  Cervical Carcinoma: number analyzed (Participants) | 13
  Cervical Carcinoma | 7.7 [0.2 to 36.0]
  Vaginal/Vulvar Carcinoma: number analyzed (Participants) | 12
  Vaginal/Vulvar Carcinoma | 0 [0.0 to 26.5]
  Merkel Cell Carcinoma: number analyzed (Participants) | 37
  Merkel Cell Carcinoma | 2.7 [0.1 to 14.2]

4. Primary Outcome: Metastatic: Investigator-Assessed Objective Response Rate (ORR)
Description: Objective response rate (ORR) is defined as the percentage of participants with a best overall response (BOR) of confirmed complete response (CR) or partial response (PR) using RECIST 1.1 criteria. An ORR in excess of 10% will be considered of clinical interest, and an ORR of 25% or greater will be considered of strong clinical interest.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Participants with the following diseases will be assessed:
  1. EBV positive related gastric cancer;
  2. HPV positive SCCHN;
  3. Other anogenital HPV associated cancers;
  4. GYN (Cervical, Vaginal, Vulvar) carcinoma;
  5. Merkel cell carcinoma (MCC);
  6. Nasopharyngeal carcinoma (NPC)
Time Frame: From the date of first dose to the date of the initial objectively documented tumor progression or the date of the last tumor assessment prior to subsequent therapy (Up to 65 months)
Population: All treated participants in the metastatic cohorts
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Metastatic Monotherapy | Metastatic Combo A | Metastatic Combo B | Metastatic Combo C | Metastatic Combo D
Number analyzed (Participants) | 113 | 195 | 133 | 8 | 6
Percentage of participants
  EBV positive related gastric cancer: number analyzed (Participants) | 14 | 0 | 0 | 0 | 0
  EBV positive related gastric cancer | 14.3 [1.8 to 42.8] |  |  |  |
  HPV positive SCCHN: number analyzed (Participants) | 26 | 42 | 0 | 8 | 0
  HPV positive SCCHN | 11.5 [2.4 to 30.2] | 31.0 [17.6 to 47.1] |  | 0 [0.0 to 36.9] |
  Other anogenital HPV associated cancers: number analyzed (Participants) | 0 | 23 | 21 | 0 | 0
  Other anogenital HPV associated cancers |  | 34.8 [16.4 to 57.3] | 28.6 [11.3 to 52.2] |  |
  SCCHN I-O naive: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6
  SCCHN I-O naive |  |  |  |  | 16.7 [0.4 to 64.1]
  Cervical: number analyzed (Participants) | 19 | 45 | 45 | 0 | 0
  Cervical | 26.3 [9.1 to 51.2] | 31.1 [18.2 to 46.6] | 40.0 [25.7 to 55.7] |  |
  Cervical first line: number analyzed (Participants) | 0 | 0 | 44 | 0 | 0
  Cervical first line |  |  | 36.4 [22.4 to 52.2] |  |
  Cervical second line: number analyzed (Participants) | 0 | 0 | 23 | 0 | 0
  Cervical second line |  |  | 39.1 [19.7 to 61.5] |  |
  Vaginal/Vulvar: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0
  Vaginal/Vulvar | 20.0 [0.5 to 71.6] |  |  |  |
  MCC: number analyzed (Participants) | 25 | 43 | 0 | 0 | 0
  MCC | 64.0 [42.5 to 82.0] | 58.1 [42.1 to 73.0] |  |  |
  NPC: number analyzed (Participants) | 24 | 42 | 0 | 0 | 0
  NPC | 16.7 [4.7 to 37.4] | 26.2 [13.9 to 42.0] |  |  |

5. Secondary Outcome: Metastatic: Investigator-Assessed Duration of Response (DoR)
Description: Duration of response (DoR) is defined as the time from first confirmed response (complete response or partial response) to the date of the initial objectively documented tumor progression as determined per investigator assessment using RECIST 1.1 criteria or death due to any cause, whichever occurs first. Participants with the following diseases will be assessed:
  1. EBV positive related gastric cancer;
  2. HPV positive SCCHN;
  3. Other anogenital HPV associated cancers;
  4. GYN (Cervical, Vaginal, Vulvar) carcinoma;
  5. Merkel cell carcinoma (MCC);
  6. Nasopharyngeal carcinoma (NPC) NOTE: "Cervical, Randomized" and "Cervical, Pooled" are not mutually exclusive categories.
Time Frame: From first confirmed response (complete response or partial response) to the date of the initial objectively documented tumor progression or death due to any cause, whichever occurs first (Up to 83 months)
Population: All complete and partial responders in the metastatic cohorts
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Metastatic Monotherapy | Metastatic Combo A | Metastatic Combo B | Metastatic Combo C | Metastatic Combo D
Number analyzed (Participants) | 30 | 72 | 50 | 0 | 1
Months
  EBV positive related gastric cancer: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  EBV positive related gastric cancer | NA [NA to NA] — Median not reached as insufficient progression events among responders |  |  |  |
  HPV positive SCCHN: number analyzed (Participants) | 3 | 13 | 0 | 0 | 0
  HPV positive SCCHN | 44.25 [24.90 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold | 34.46 [10.45 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold |  |  |
  Other anogenital HPV associated cancers: number analyzed (Participants) | 0 | 8 | 5 | 0 | 0
  Other anogenital HPV associated cancers |  | 18.23 [3.68 to 27.93] | 3.71 [3.58 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold |  |
  SCCHN I-O naive: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  SCCHN I-O naive |  |  |  |  | NA [NA to NA] — Median not reached as insufficient progression events among responders
  Cervical, Randomized: number analyzed (Participants) | 5 | 14 | 18 | 0 | 0
  Cervical, Randomized | NA [35.29 to NA] — Median not reached as insufficient progression events among responders and Upper limit not calculable as upper CI bound does not cross 50% threshold | NA [8.67 to NA] — Median not reached as insufficient progression events among responders and Upper limit not calculable as upper CI bound does not cross 50% threshold | 34.07 [15.28 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold |  |
  Cervical, Pooled: number analyzed (Participants) | 0 | 0 | 45 | 0 | 0
  Cervical, Pooled |  |  | 34.07 [15.28 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold |  |
  Vaginal/Vulvar: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Vaginal/Vulvar | 4.96 [NA to NA] — Lower limit and Upper limit not calculable as upper CI bound does not cross 50% threshold |  |  |  |
  MCC: number analyzed (Participants) | 15 | 25 | 0 | 0 | 0
  MCC | 60.62 [16.72 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold | 25.86 [10.38 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold |  |  |
  NPC: number analyzed (Participants) | 4 | 12 | 0 | 0 | 0
  NPC | 9.46 [3.68 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold | 19.63 [5.55 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold |  |  |

6. Secondary Outcome: Metastatic: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from first dosing date to the date of death. A participant who has not died will be censored at last known date alive. Participants with the following diseases will be assessed:
  1. EBV positive related gastric cancer;
  2. HPV positive SCCHN;
  3. Other anogenital HPV associated cancers;
  4. GYN (Cervical, Vaginal, Vulvar) carcinoma;
  5. Merkel cell carcinoma (MCC);
  6. Nasopharyngeal carcinoma (NPC) Note: "Cervical, Randomized" and "Cervical, Pooled" are not mutually exclusive categories
Time Frame: From the first dosing date to the date of death (Up to 83 months)
Population: All treated participants in the metastatic cohorts
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Metastatic Monotherapy | Metastatic Combo A | Metastatic Combo B | Metastatic Combo C | Metastatic Combo D
Number analyzed (Participants) | 113 | 195 | 133 | 8 | 6
Months
  EBV positive related gastric cancer: number analyzed (Participants) | 14 | 0 | 0 | 0 | 0
  EBV positive related gastric cancer | 9.99 [3.09 to 30.13] |  |  |  |
  HPV positive SCCHN: number analyzed (Participants) | 26 | 42 | 0 | 8 | 0
  HPV positive SCCHN | 20.44 [13.90 to 36.50] | 17.08 [9.49 to 26.78] |  | 8.84 [2.50 to 35.06] |
  Other anogenital HPV associated cancers: number analyzed (Participants) | 0 | 23 | 21 | 0 | 0
  Other anogenital HPV associated cancers |  | 12.12 [6.83 to 29.54] | 14.06 [4.37 to 30.59] |  |
  SCCHN I-O naive: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6
  SCCHN I-O naive |  |  |  |  | 4.21 [1.68 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold
  Cervical, Randomized: number analyzed (Participants) | 19 | 45 | 45 | 0 | 0
  Cervical, Randomized | 21.55 [8.25 to 44.85] | 17.12 [10.22 to 34.79] | 22.74 [14.62 to 32.82] |  |
  Cervical, Pooled: number analyzed (Participants) | 0 | 0 | 112 | 0 | 0
  Cervical, Pooled |  |  | 20.93 [14.39 to 29.04] |  |
  Vaginal/Vulvar: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0
  Vaginal/Vulvar | 10.28 [3.88 to 23.72] |  |  |  |
  MCC: number analyzed (Participants) | 25 | 43 | 0 | 0 | 0
  MCC | 80.66 [23.26 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold | 29.83 [8.51 to 48.33] |  |  |
  NPC: number analyzed (Participants) | 24 | 42 | 0 | 0 | 0
  NPC | 22.74 [12.62 to 35.29] | 23.66 [16.82 to 41.43] |  |  |

7. Secondary Outcome: Metastatic: Investigator-Assessed Progression-Free Survival (PFS)
Description: Investigator-assessed progression free survival (PFS) is defined as the time from first dosing date to the date of the first documented tumor progression, as determined by investigators (per RECIST 1.1), or death due to any cause, whichever occurs first. Participants with the following diseases will be assessed:
  1. EBV positive related gastric cancer;
  2. HPV positive SCCHN;
  3. Other anogenital HPV associated cancers;
  4. GYN (Cervical, Vaginal, Vulvar) carcinoma;
  5. Merkel cell carcinoma (MCC);
  6. Nasopharyngeal carcinoma (NPC) Note: "Cervical, Randomized" and "Cervical, Pooled" are not mutually exclusive categories
Time Frame: From the first dosing date to the date of the first documented tumor progression or death due to any cause, whichever occurs first (Up to 83 months)
Population: All treated participants in the metastatic cohorts
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Metastatic Monotherapy | Metastatic Combo A | Metastatic Combo B | Metastatic Combo C | Metastatic Combo D
Number analyzed (Participants) | 113 | 195 | 133 | 8 | 6
Months
  EBV positive related gastric cancer: number analyzed (Participants) | 14 | 0 | 0 | 0 | 0
  EBV positive related gastric cancer | 2.94 [1.05 to 3.75] |  |  |  |
  HPV positive SCCHN: number analyzed (Participants) | 26 | 42 | 0 | 8 | 0
  HPV positive SCCHN | 3.25 [1.84 to 6.93] | 3.71 [1.77 to 6.80] |  | 3.81 [1.77 to 7.39] |
  Other anogenital HPV associated cancers: number analyzed (Participants) | 0 | 23 | 21 | 0 | 0
  Other anogenital HPV associated cancers |  | 4.63 [1.94 to 14.29] | 3.58 [2.04 to 7.49] |  |
  SCCHN I-O naive: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6
  SCCHN I-O naive |  |  |  |  | 1.81 [1.08 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold
  Cervical, Randomized: number analyzed (Participants) | 19 | 45 | 45 | 0 | 0
  Cervical, Randomized | 5.09 [1.87 to 9.07] | 3.75 [3.32 to 9.23] | 7.11 [3.71 to 17.25] |  |
  Cervical, Pooled: number analyzed (Participants) | 0 | 0 | 112 | 0 | 0
  Cervical, Pooled |  |  | 5.85 [3.75 to 9.03] |  |
  Vaginal/Vulvar: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0
  Vaginal/Vulvar | 3.75 [1.22 to 8.15] |  |  |  |
  MCC: number analyzed (Participants) | 25 | 43 | 0 | 0 | 0
  MCC | 21.32 [9.20 to 62.52] | 8.39 [3.71 to 24.34] |  |  |
  NPC: number analyzed (Participants) | 24 | 42 | 0 | 0 | 0
  NPC | 1.94 [1.54 to 3.58] | 5.36 [2.37 to 9.23] |  |  |

8. Post Hoc Outcome: Metastatic: Investigator-Assessed Objective Response Rate (ORR) Extended Collection
Description: ORR is defined as the percentage of participants with a best overall response (BOR) of confirmed complete response (CR) or partial response (PR) using RECIST 1.1 criteria. An ORR in excess of 10% will be considered of clinical interest, and an ORR of 25% or greater will be considered of strong clinical interest.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Participants with the following diseases will be assessed:
  1. EBV positive related gastric cancer;
  2. HPV positive SCCHN;
  3. Other anogenital HPV associated cancers;
  4. GYN (Cervical, Vaginal, Vulvar) carcinoma;
  5. Merkel cell carcinoma (MCC);
  6. Nasopharyngeal carcinoma (NPC) Note: "Cervical, Randomized" and "Cervical, Pooled" are not mutually exclusive categories
Time Frame: From the date of first dose to the date of the initial objectively documented tumor progression or the date of the last tumor assessment prior to subsequent therapy (Up to 83 months)
Population: All treated participants in the metastatic cohorts
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Metastatic Monotherapy | Metastatic Combo A | Metastatic Combo B | Metastatic Combo C | Metastatic Combo D
Number analyzed (Participants) | 113 | 195 | 133 | 8 | 6
Percentage of participants
  EBV positive related gastric cancer: number analyzed (Participants) | 14 | 0 | 0 | 0 | 0
  EBV positive related gastric cancer | 14.3 [1.8 to 42.8] |  |  |  |
  HPV positive SCCHN: number analyzed (Participants) | 26 | 42 | 0 | 8 | 0
  HPV positive SCCHN | 11.5 [2.4 to 30.2] | 31.0 [17.6 to 47.1] |  | 0 [0.0 to 36.9] |
  Other anogenital HPV associated cancers: number analyzed (Participants) | 0 | 23 | 21 | 0 | 0
  Other anogenital HPV associated cancers |  | 34.8 [16.4 to 57.3] | 23.8 [8.2 to 47.2] |  |
  SCCHN I-O naive: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6
  SCCHN I-O naive |  |  |  |  | 16.7 [0.4 to 64.1]
  Cervical, Randomized: number analyzed (Participants) | 19 | 45 | 45 | 0 | 0
  Cervical, Randomized | 26.3 [9.1 to 51.2] | 31.1 [18.2 to 46.6] | 40.0 [25.7 to 55.7] |  |
  Cervical, Pooled: number analyzed (Participants) | 0 | 0 | 112 | 0 | 0
  Cervical, Pooled |  |  | 40.2 [31.0 to 49.9] |  |
  Vaginal/Vulvar: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0
  Vaginal/Vulvar | 20.0 [0.5 to 71.6] |  |  |  |
  MCC: number analyzed (Participants) | 25 | 43 | 0 | 0 | 0
  MCC | 60.0 [38.7 to 78.9] | 58.1 [42.1 to 73.0] |  |  |
  NPC: number analyzed (Participants) | 24 | 42 | 0 | 0 | 0
  NPC | 16.7 [4.7 to 37.4] | 28.6 [15.7 to 44.6] |  |  |

ADVERSE EVENTS:
Time Frame: SAEs and Other AEs are assessed from first dose to 100 days post last dose (Up to 83 months) Participants were assessed for all-cause mortality from their first dose to their study completion (Up to 84 months)
Groups:
- Neoadjuvant: Nivolumab IV over 30 minutes at 240 mg for 2 doses, on Day 1 and Day 15
Arm/Group | Metastatic Monotherapy | Metastatic Combo A | Metastatic Combo B | Metastatic Combo C | Metastatic Combo D | Neoadjuvant
All-Cause Mortality (participants affected / at risk) | 82/113 | 133/195 | 86/133 | 7/8 | 5/6 | 40/123
Serious Adverse Events (participants affected / at risk) | 59/113 | 130/195 | 99/133 | 5/8 | 5/6 | 40/123
Other Adverse Events (participants affected / at risk) | 110/113 | 189/195 | 129/133 | 7/8 | 5/6 | 108/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metastatic Monotherapy (N=113) | Metastatic Combo A (N=195) | Metastatic Combo B (N=133) | Metastatic Combo C (N=8) | Metastatic Combo D (N=6) | Neoadjuvant (N=123)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 5 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 0 | 0 | 0 | 0
Autoimmune pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 2 | 2 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 4 | 0 | 0 | 0 | 0
Glucocorticoid deficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 1 | 0 | 0 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 3 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thyroid disorder (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 2 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anorectal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 3 | 11 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 9 | 4 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 1 | 3 | 0 | 0 | 1
Immune-mediated pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 7 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 1
Oesophageal motility disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4 | 2 | 0 | 0 | 1
Asthenia (General disorders) | 1 | 1 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Complication associated with device (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 1 | 2 | 1 | 0 | 0 | 0
Disease progression (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 0 | 1
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperthermia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 3
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 2 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 2 | 0 | 0 | 0 | 1
Performance status decreased (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 5 | 7 | 0 | 0 | 2
Sudden death (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Autoimmune cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 3 | 0 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gallbladder rupture (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 6 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 3 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abscess neck (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Clostridial sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Device related sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Large intestine infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0
Medical device site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Meningitis aseptic (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Periorbital infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 3 | 1 | 0 | 1 | 0
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 1 | 4 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 3 | 6 | 4 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 11 | 7 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0
Recall phenomenon (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood pressure decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
General physical condition abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 2 | 2 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Respiratory syncytial virus test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 4 | 2 | 0 | 0 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 4 | 1 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24 | 39 | 21 | 2 | 3 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0
Tumour obstruction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0
Basal ganglia infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bell's palsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Carotid artery aneurysm (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Monoparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 3 | 0 | 0 | 0 | 1
Device occlusion (Product Issues) | 1 | 2 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 3 | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 5 | 8 | 0 | 0 | 0
Autoimmune nephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 2 | 2 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 3 | 0 | 0 | 0 | 0
Renal haematoma (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 2 | 1 | 0 | 0 | 0
Urogenital fistula (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1 | 2 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0 | 1
Vulval disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0 | 2 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 10 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Debridement (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Arterial haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 2 | 1 | 1 | 0 | 1 | 0
Iliac vein stenosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metastatic Monotherapy (N=113) | Metastatic Combo A (N=195) | Metastatic Combo B (N=133) | Metastatic Combo C (N=8) | Metastatic Combo D (N=6) | Neoadjuvant (N=123)
Anaemia (Blood and lymphatic system disorders) | 28 | 53 | 42 | 2 | 2 | 11
Ear pain (Ear and labyrinth disorders) | 3 | 4 | 1 | 0 | 1 | 2
Vertigo (Ear and labyrinth disorders) | 6 | 1 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 9 | 21 | 0 | 0 | 4
Hypothyroidism (Endocrine disorders) | 17 | 39 | 31 | 2 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 18 | 28 | 30 | 1 | 0 | 8
Abdominal pain upper (Gastrointestinal disorders) | 12 | 9 | 5 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 6 | 7 | 0 | 0 | 4
Constipation (Gastrointestinal disorders) | 27 | 51 | 37 | 1 | 0 | 21
Diarrhoea (Gastrointestinal disorders) | 31 | 61 | 54 | 1 | 2 | 22
Dry mouth (Gastrointestinal disorders) | 8 | 13 | 6 | 1 | 0 | 6
Dyspepsia (Gastrointestinal disorders) | 4 | 11 | 7 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 10 | 12 | 2 | 4 | 0 | 21
Nausea (Gastrointestinal disorders) | 25 | 45 | 48 | 2 | 3 | 42
Stomatitis (Gastrointestinal disorders) | 7 | 5 | 4 | 0 | 0 | 5
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 21 | 31 | 33 | 1 | 0 | 14
Asthenia (General disorders) | 18 | 26 | 23 | 0 | 0 | 11
Chest pain (General disorders) | 6 | 2 | 1 | 1 | 0 | 0
Chills (General disorders) | 6 | 10 | 9 | 0 | 0 | 3
Face oedema (General disorders) | 2 | 6 | 1 | 0 | 1 | 3
Facial pain (General disorders) | 3 | 0 | 0 | 0 | 1 | 3
Fatigue (General disorders) | 47 | 81 | 46 | 6 | 1 | 40
Gait disturbance (General disorders) | 0 | 2 | 1 | 0 | 1 | 0
Inflammation (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 4 | 12 | 2 | 0 | 0 | 3
Localised oedema (General disorders) | 0 | 2 | 0 | 0 | 0 | 8
Malaise (General disorders) | 4 | 3 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 4 | 6 | 5 | 0 | 0 | 15
Non-cardiac chest pain (General disorders) | 5 | 3 | 3 | 1 | 0 | 2
Oedema peripheral (General disorders) | 16 | 21 | 20 | 1 | 2 | 6
Pain (General disorders) | 3 | 9 | 4 | 1 | 1 | 2
Pyrexia (General disorders) | 14 | 34 | 33 | 0 | 2 | 13
Bronchitis (Infections and infestations) | 8 | 3 | 1 | 0 | 0 | 1
Candida infection (Infections and infestations) | 3 | 5 | 0 | 1 | 0 | 3
Conjunctivitis (Infections and infestations) | 6 | 4 | 3 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Mucosal infection (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 10 | 14 | 3 | 0 | 0 | 0
Oral bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 3 | 7 | 2 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 6 | 4 | 3 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 7 | 27 | 8 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 9 | 21 | 31 | 0 | 0 | 9
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 11 | 4 | 0 | 0 | 4
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 3 | 3 | 0 | 0 | 0 | 9
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 15
Alanine aminotransferase increased (Investigations) | 8 | 26 | 22 | 0 | 0 | 4
Amylase increased (Investigations) | 6 | 20 | 12 | 1 | 0 | 7
Aspartate aminotransferase increased (Investigations) | 10 | 25 | 20 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 5 | 10 | 7 | 0 | 0 | 3
Blood creatinine increased (Investigations) | 11 | 19 | 13 | 0 | 0 | 4
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Lipase increased (Investigations) | 17 | 27 | 17 | 2 | 0 | 7
Lymphocyte count decreased (Investigations) | 1 | 16 | 3 | 0 | 0 | 2
Platelet count decreased (Investigations) | 0 | 11 | 0 | 0 | 0 | 1
Troponin increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 10 | 24 | 8 | 2 | 0 | 15
White blood cell count decreased (Investigations) | 2 | 10 | 4 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 24 | 48 | 32 | 2 | 1 | 15
Dehydration (Metabolism and nutrition disorders) | 1 | 9 | 3 | 0 | 0 | 8
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 9 | 4 | 0 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 16 | 9 | 0 | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 14 | 16 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 20 | 15 | 1 | 0 | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 | 14 | 17 | 1 | 0 | 10
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 24 | 14 | 1 | 1 | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 20 | 3 | 1 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 35 | 26 | 2 | 1 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 28 | 19 | 1 | 1 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 6 | 7 | 7 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 10 | 4 | 1 | 0 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8 | 11 | 2 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 2 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 19 | 10 | 0 | 0 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 7 | 1 | 1 | 0 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 13 | 9 | 0 | 0 | 4
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 5 | 3 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 12 | 19 | 15 | 0 | 0 | 6
Dysgeusia (Nervous system disorders) | 7 | 3 | 3 | 0 | 0 | 10
Headache (Nervous system disorders) | 13 | 31 | 22 | 0 | 2 | 6
Paraesthesia (Nervous system disorders) | 2 | 3 | 2 | 2 | 0 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 4 | 4 | 0 | 1 | 8
Anxiety (Psychiatric disorders) | 10 | 8 | 4 | 1 | 0 | 9
Confusional state (Psychiatric disorders) | 1 | 5 | 2 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 10 | 23 | 8 | 1 | 1 | 2
Pelvic pain (Reproductive system and breast disorders) | 2 | 6 | 7 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 6 | 7 | 0 | 0 | 4
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 0 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 49 | 17 | 2 | 1 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 30 | 13 | 2 | 1 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 1 | 0 | 0 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 11 | 4 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 10 | 3 | 0 | 1 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 1 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 9 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 7 | 0 | 0 | 3
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 1 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 14 | 12 | 0 | 1 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 23 | 60 | 35 | 0 | 1 | 11
Rash (Skin and subcutaneous tissue disorders) | 17 | 49 | 16 | 1 | 0 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 | 20 | 25 | 0 | 0 | 6
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 2 | 0
Haematoma (Vascular disorders) | 2 | 2 | 0 | 1 | 0 | 2
Hypertension (Vascular disorders) | 10 | 7 | 5 | 1 | 0 | 12
Hypotension (Vascular disorders) | 5 | 10 | 4 | 0 | 1 | 4
Lymphoedema (Vascular disorders) | 4 | 4 | 5 | 1 | 1 | 2
Venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT02488759/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT02488759/SAP_001.pdf